CLINICAL TRIAL: NCT04076137
Title: Clinical Study of Targeted T-cell Therapy in Solid Tumors
Brief Title: Targeted T-cell Therapy in Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benhealth Biopharmaceutical (Shenzhen) Co., Ltd. (Industry)
Collaborators: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BK2019.01
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Malignant Solid Tumor
Keywords: Targeted T-cell; HER2; MUC1; CEA; EGFR; GPC3
MeSH Terms: interventions — Antibodies, Bispecific; Decitabine

STUDY DESIGN:
Intervention Model Description: This is a single-center, open, single-arm controlled prospective clinical study to investigate the efficacy and safety of targeted T-cell therapy in solid tumors.
Masking Description: targeted activated T-cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted T-cell (Experimental): This study is a pre-phase I immunotherapy trial in 10 people with malignant solid tumor consisting of 9 infusions of bispecific antibody armed anti-CD3-Actibated T cells(ATC) to determine safety, maximum tolerated dose (MTD), technical feasibility, immune responses.
  Interventions: Other: Targeted T-cell armed with bispecific antibody (Decitabine)

INTERVENTIONS:
Other: Targeted T-cell armed with bispecific antibody (Decitabine) — In this study, 10 patients eligible for the study were clinically screened for intravenous infusion of targeted activated T cells,every participant has a unique identification number and emergency letter which have the information of group.
  Other Names: decitabine

SUMMARY:
This is a single-center, open, single-arm controlled prospective clinical trial of patients with solid tumors treated with targeted activation of T cells through intravenous infusion.The purpose of this study was to evaluate the clinical efficacy and safety of targeted activated T cells in the treatment of solid tumors.

DETAILED DESCRIPTION:
In China, malignant tumors have become the leading cause of death for urban and rural residents, with solid tumors accounting for 77 percent.Immunotherapy is considered one of the most promising ways to fight cancer.This study is a single-center, open, single-arm controlled clinical trial (after intravenous infusion of targeted T cells, compare the changes of self-lesion). The essence of this study is to collect immune cells to the surrounding of tumor cells, so that immune cells can kill tumor cells at close range.The researchers plan to enroll 10 patients with solid tumors and follow them up to the end of the study after completing 9 courses of treatment.The results of this study were statistically analyzed using RECIST1.1 records.

ELIGIBILITY:
Inclusion Criteria:1. Age: 18~75 years old; 2. Patients with solid tumors still show progress after radiotherapy, chemotherapy and targeted therapy, with at least one measurable lesion; 3. No congenital autoimmune diseases or immunodeficiency diseases;' 4. At least one or more solid tumor targets of HER2, MUC1, CEA, EGFR and GPC3 were positive by immunohistochemical examination of tumor tissues; 5. No serious infectious diseases (hepatitis b, c, syphilis, AIDS); 6. Sign informed consent voluntarily. -

Exclusion Criteria:1. The researchers determined that the patient could not complete 6 courses of treatment.

2. Patients with t-cell lymphoma. 3. Pregnant or lactating female patients, or those who do not want to use contraception during the trial.

4. Allergic to both CT and MRI contrast agents and unable to conduct imaging evaluation.

5. Other patients in the treated group who were considered as unfit for cell therapy.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
OS | 1 year .
  Overrall survival.The time of patient from randomization to death caused by any cause.

SECONDARY OUTCOMES:
PFS | 1 year.
  Progression-free survival.The time of patients from randomization to death caused by the progression of the tumor or any cause.

OTHER OUTCOMES:
TTP | 1 year.
  Time tumor progression.The time of patient from randomization to objective progress of the tumor.
DCR | 1 year.
  Disease control rate.The proportion of patients who had a best response rating of complete response, partial response, or stable disease.
ORR | 1 year.
  Objective response rate.The proportion of patients who had a best response rating of complete response and partial response.
SRR | 1 year.
  Symptom remission rate. The proportion of symptoms are alleviated in all evaluative cases.

CONTACTS AND LOCATIONS:
Overall Officials: Zeqiang Zhou, Doctor, Study Chair — Department of oncology, the second people's hospital of shenzhen; Wenli Liang, Doctor, Study Director — Department of oncology, the second people's hospital of shenzhen; Liang Xiao, Doctor, Principal Investigator — Department of oncology, the second people's hospital of shenzhen; Lin Lin, Doctor, Principal Investigator — Department of oncology, the second people's hospital of shenzhen; Meixiang Li, Doctor, Principal Investigator — Department of oncology, the second people's hospital of shenzhen
Locations (1):
- Department of oncology, the second people's hospital of shenzhen, Shenzhen, Guangdong, China